CLINICAL TRIAL: NCT07029945
Title: A Phase 1/2 Study of the Safety and Efficacy of BRX011 Oral Administration Once Daily in Subjects With Geographic Atrophy Secondary to Age-Related Macular Degeneration
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biojiva LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BRX011-001
Record Dates: First submitted 2025-06-12; First posted 2025-06-19 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Geographic Atrophy
Keywords: Geographic Atrophy; AMD; Age-Related Macular Degeneration; Oral; Oral Therapy; GA
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BRX011 (Active Comparator)
  Interventions: Drug: BRX011
- Safflower Oil (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BRX011 — Subjects will ingest BRX011 orally, as capsules.
  Arms: BRX011
Drug: Placebo — Subjects will ingest Placebo orally, as capsules.
  Arms: Safflower Oil

SUMMARY:
This study aims to evaluate the safety and efficacy of BRX011, an oral medication, taken once daily by participants with geographic atrophy secondary to age-related macular degeneration. The study is conducted in phases 1 and 2, focusing on assessing both safety (tolerability) and effectiveness (efficacy) of the treatment.

Participants: Adults with geographic atrophy due to age-related macular degeneration.

Treatment: BRX011 or Placebo is taken once daily as per the protocol.

Duration: The study involves multiple visits over 96 weeks to monitor participants' health and response to treatment.

Safety Monitoring: Regular checks for adverse events and health status to ensure participant well-being. Checks will include examination of vital signs, clinical labs, ocular exams, and ocular imaging.

Primary Outcome Measure: Efficacy of BRX011 in the annual rate of change in the square root of GA area, as specified in the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥55 years
2. Visual acuity in the study eye at Screening/Baseline

   1. BCVA ≥35 letters using ETDRS charts (≥20/200 Snellen equivalent)
   2. LLD >5 letters
3. Clinical diagnosis of GA secondary to AMD. CNV in the fellow eye is permitted.

(5) Clarity of ocular media, adequate pupillary dilation, and fixation to permit the evaluation of the eye, as determined by the investigator

(6) Female subjects must be of non-child-bearing potential (WONCBP), defined as:

(a) A woman who had surgical sterilization (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy) (b) A woman ≥ 60 years of age (c) A woman ≥ 55 and < 60 years of age who fulfills at least one of the following: (i) A cessation of menses for at least 12 months and a folliclestimulating hormone (FSH) test confirming non-childbearing potential (refer to laboratory reference ranges for confirmatory levels) (ii) A cessation of menses for at least 24 months without FSH levels confirmed.

(7) Willing and able to give informed consent and to comply with the study procedures and assessments

Exclusion Criteria:

1. GA secondary to a condition other than AMD such as Stargardt disease, cone rod dystrophy or toxic maculopathies like plaquenil maculopathy in either eye
2. Any history documented or active CNV
3. Any ocular condition other than GA secondary to AMD that may require surgery or medical intervention during the study period

(5) History of vitrectomy surgery, submacular surgery, other surgical intervention for AMD, corneal transplant, glaucoma filtration surgery, or cataract surgery within 3 months prior to Screening/Baseline

(6) History of intravitreal injection of anti-vascular endothelial growth factor (VEGF) therapies in the study eye at any time, history of intravitreal injection of any agent (e.g., triamcinolone) in the study eye within the last 3 months prior to study enrollment. A single intraoperative administration of a corticosteroid during cataract surgery at least 3 months prior to Screening is permitted

(7) History of laser therapy in the macular region in the study eye, prior treatment with photobiomodulation, external-beam radiation therapy or transpupillary thermotherapy in study eye

(8) Previous cell-based intraocular treatment in the study eye or previous expression vector-mediated intraocular treatments in either eye (i.e., gene therapy), any previous treatment with any deuterated molecules for eye diseases (e.g., deuterated vitamin A)

(9) History of idiopathic or autoimmune-associated uveitis, ocular or intraocular conditions, and infectious or inflammatory ocular disease. Active uveitis and infectious conjunctivitis, keratitis, scleritis or endophthalmitis

(11) Active malignancy within the previous 12 months except for appropriately treated carcinoma in situ of cervix, resolved non-melanoma skin carcinoma, and prostate cancer with a Gleason score of less than or equal to (≤) 6, and a stable prostate-specific antigen for greater than or equal to (≥) 12 months

(13) Intake of omega-3 supplements (e.g., fish oil, cod liver oil, krill oil, edible algae oil, flax oil) or prescription omega-3 drugs (e.g., Lovaza® , Vascepa® , Epanova® ) in the past 4 weeks prior to Screening and throughout the duration of the study; intake of supplements containing Lutein, zeaxanthin and or mesozeaxanthin (e.g., Ocuvite® , PreserVision® , SYSTANE ICAPS ® or other AREDS supplements) in the past 4 weeks prior to Screening and throughout the duration of the study

(14) Participation in an interventional clinical study within the past 30 days of Screening, or interventional GA studies within the past 5 months prior to Screening

(15) Treatment with SYFOVRE ®or IZERVAY ®within 3 months prior to Screening

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-07-07 (Estimated); Primary Completion 2026-11-11 (Estimated); Study Completion 2027-02-11 (Estimated)

PRIMARY OUTCOMES:
Annual rate of change in the square root of GA area | Baseline (Day 0) to Week 96
  Annual rate of change in the square root of GA area assessed by FAF

SECONDARY OUTCOMES:
Change in low luminance deficit | Baseline (Day 0) to Week 96
Change in ETDRS BCVA | Baseline (Day 0) to Week 96